CLINICAL TRIAL: NCT04447950
Title: A Randomized, Double Blind, Placebo Controlled Evaluation Trial of the Benefit in Quadratus Lumborum Block as a Postoperative Analgesic Technique for a Lumbar Spine Decompression and Fusion Surgery
Brief Title: Randomized Control Trial of Quadratus Lumborum Block for Lumbar Spine Decompression and Fusion Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Ely Ashkenazy, Dr Ely Ashkenazy, neurosurgeon, Assuta Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0012-20
Record Dates: First submitted 2020-06-20; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Spinal Stenosis Lumbar; Spondylolisthesis; Fusion of Spine, Lumbar Region; Degeneration Spine
MeSH Terms: conditions — Spondylolisthesis | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 2 arms of a RCT.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Rotating nurse assigning the arm, scrubbed nurse preparing syringe for injection with a clear liquid - saline vs saline and Marcaine, surgeon blinded to type of liquid in syringe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Posterior QL block with 20-40 cc of Bupivocaine in posterior border of Quadratum Lumborum muscle at the end of the operation.
  Interventions: Procedure: Type 2/posterior Quadratus Lumborum block
- Placebo group (Placebo Comparator): Posterior QL block with 40 cc of Saline in posterior border of Quadratum Lumborum muscle at the end of the operation.
  Interventions: Procedure: Placebo block with Saline

INTERVENTIONS:
Procedure: Type 2/posterior Quadratus Lumborum block — Injection of local anaesthetic into posterior boundry of Quadratus Lumborum muscle.
  Arms: Study group
Procedure: Placebo block with Saline — Injection of saline into posterior boundary of Quadratus Lumborum muscle.
  Arms: Placebo group

SUMMARY:
Lumbar spinal decompression and fusion is a commonly performed procedure fro neural impingement and back pain from a variety of pathologies. The importance of pain control in the postoperative period for spinal surgery has been discussed and proven extensively, with both immediate and delayed reduction in complications and improved clinical results.

Quadratus lumborum (QL) block was introduced in 2007 and is performed under ultrasound guidance for perioperative pain management in various surgeries.However, the plane for a posterior QL block can be easily reached during open midline spinal surgery.

The investigators hypothesize that the posterior QL block is an effective analgesic tool for lumbar laminectomy surgery, because in lumbar laminectomy the quadratus lumborum is already exposed and is in direct visual contact. For that reason it is imperative to test the benefits of this procedure.

This is a double blinded randomized control study to assess the results of intra-operative QL block performed for lumbar decompression and fusion.

DETAILED DESCRIPTION:
Spinal decompression is a surgical procedure that is performed to alleviate pain caused by pinched nerves (neural impingement). Surgical options for decompressing the lumbar spine vary from minimally invasive disc decompression to open laminectomy and foraminotomy. The lumbar spine decompression and fusion differs from a microdiscectomy in that the incision is longer and there is more muscle stripping. Lumbar spinal decompression is a commonly performed procedure and the conventional open techniques of decompression remain the gold standard of treatment.

During a lumbar decompression back surgery, a small portion of the bone over the nerve root and/or disc material from under the nerve root is removed to give the nerve root more space and provide a better healing environment. A lumbar spine decompression and fusion is typically performed to relieve the lumbar spinal stenosis symptoms. The goal of the surgery is to allow more space for the nerve root, thus reducing pain (and potentially any leg weakness or neurological symptoms) and restoring the patient's ability to participate in everyday activities[1].

Quadratus lumborum (QL) block was introduced in 2007 and is performed for perioperative pain management in various abdominal, pelvic, gynecological and hip procedures in all age groups[2]. Four types of QL block were described, differentiated by the exact location of the anesthetic injection. Type 1/lateral QL block is performed at the lateral border of the QL muscle, type 2/posterior QL block is performed at the medial edge of the QL muscle (at the border or the spine erector muscles and the thoraco-lumbar fascia), type 3/anterior is performed between the QL muscle and the psoas major and type 4 is intramuscular (see figure 1). In the majority of cases, these blocks are performed pre/post operatively under ultrasound guidance. There are sporadic reports of QL block performed for lumbar spinal surgery [3, 4].However, the plane for a type 2 QL block can be easily reached during open midline spinal surgery.

The importance of pain control in the postoperative period for spinal surgery has been discussed and proven extensively, with both immediate and delayed reduction in complications and improved clinical results [5, 6].

The investigators hypothesize that the type 2 QL block is an effective analgesic tool for lumbar laminectomy surgery, because in lumbar laminectomy the quadratus lumborum is already exposed and is in direct visual contact. For that reason it is imperative, in our opinion, to test its benefits of this procedure.

Study's objective:

To test the safety and efficacy of open quadratus lumborum block as an add-on postoperative analgesic technique for lumbar spine decompression and fusion.

Study design:

This is a pilot comparative study, double blind and placebo controlled . Patients scheduled for a lumbar spine decompression and fusion will be divided randomly into two groups of N=50 each. Subjects in both groups will receive an intra-operative exposure of the posterior QL block plane, with injection of long acting local anesthetic for group A and Saline for group B. Both groups will be monitored during their admission in the department for opioid dose administered, reported pain levels (NRS), narcotics side effects (delirium, urinary retention, falls) and general operative complications. Patient pain levels, satisfaction and general complications will be gathered during clinic follow up.

Methods:

Patients arriving to undergo lumbar spine decompression and fusion will be offered to participate in the study. They will receive a thorough explanation about the study and will sign an informed consent form. The division into each group will be done randomly on a one by one basis, by an operating room nurse. The scrubbed nurse will be exposed to the nature of the substance injected for its sterile preparation, however the surgeons will be blinded to it. Patients will be blinded to their study arm until the end of the study. The lumbar laminectomy (open decompression) procedure will be performed as usual:

* First, the back is approached through a two-inch to five-inch long incision in the midline of the back, and the left and right back muscles (erector spinae) are dissected off the lamina on both sides and at multiple levels.
* After the spine is approached, the lamina is removed (laminectomy), allowing visualization of the nerve roots.
* The facet joints, which are directly over the nerve roots, may then be undercut (trimmed) to give the nerve roots more room.
* Fusion will be performed with pedicular screws and rods and when indicated an interbody device.

Study group A will be given an analgesic injection into the quadratus lumborum, comprising of Marcaine 0.25% with normal saline (for a total of 20 ml per side). Study group B will receive an identical procedure, however with 20 ml normal saline alone per side. Time required to perform the block for both sides will be measured.

The postoperative regime will include a standardized pain protocol as is used in routine practice. all other operative or postoperative procedures are the same for both groups. Data will be collected from nurses and physical therapy as well as discharge notes. A standardized form for obtaining data will be used in clinic follow up at 2-3 weeks and 3-4 months.

Safety data collected:

A subjective report of each patient regarding any adverse events will be collected by the study nurse during their recovery. The surgeon will report at the end of each operation if there were any adverse events and level of difficulty administrating the injection on designated forms.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at the ages of 18-80 suffering from leg + back pain or neurological claudication.
* Undergoing an elective 1-3 level lumbar laminectomy & fusion at Assuta medical center.

Exclusion Criteria:

* Chronic narcotic treatment (more than 3 months)
* Current active Infection.
* Underwent any other major operation in the last two months.
* Known hypersensitivity to local anaesthetic
* Previous lumbar instrumentation (revision of decompression to decompression with fusion will be included)
* Non Ambulatory patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in the use of post-operative narcotics | Will be reported for each postoperative day during the inpatient stay of the patient to a maximum of 7 days.
  Difference in MME (morphine milligrams equivalent) of inpatient narcotics consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Ely Ashkenazy, MD, Principal Investigator — Neurosurgeon, Assuta medical center
Locations (1):
- The Israeli spine center, Assuta medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benz RJ, Garfin SR. Current techniques of decompression of the lumbar spine. Clin Orthop Relat Res. 2001 Mar;(384):75-81. doi: 10.1097/00003086-200103000-00010. PMID 11249182
- [Background] Elsharkawy H. Quadratus Lumborum Blocks. Adv Anesth. 2017;35(1):145-157. doi: 10.1016/j.aan.2017.07.007. Epub 2017 Oct 3. No abstract available. PMID 29103570
- [Background] Iwamitsu R, Ueshima H, Otake H. RETRACTED: Intermittent bilateral posterior quadratus lumborum block was effective for pain management in lumbar spinal fusion. J Clin Anesth. 2017 Nov;42:16. doi: 10.1016/j.jclinane.2017.08.012. Epub 2017 Aug 6. No abstract available. PMID 28793274 (Retraction: PMID 35537960 J Clin Anesth. 2022 Sep;80:110818)
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experience of anterior quadratus lumborum block after lumber surgery. J Clin Anesth. 2017 Feb;37:131. doi: 10.1016/j.jclinane.2016.12.014. Epub 2017 Jan 9. No abstract available. PMID 28235503 (Retraction: PMID 35393201 J Clin Anesth. 2022 Aug;79:110740)
- [Background] Yoo JS, Ahn J, Buvanendran A, Singh K. Multimodal analgesia in pain management after spine surgery. J Spine Surg. 2019 Sep;5(Suppl 2):S154-S159. doi: 10.21037/jss.2019.05.04. PMID 31656869
- [Background] Pugely AJ, Martin CT, Gao Y, Mendoza-Lattes S. Causes and risk factors for 30-day unplanned readmissions after lumbar spine surgery. Spine (Phila Pa 1976). 2014 Apr 20;39(9):761-8. doi: 10.1097/BRS.0000000000000270. PMID 24525993
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269